CLINICAL TRIAL: NCT06103214
Title: The Effects of Two Hemodilution Methods on Vascular Endothelial Function in Patients Undergoing Primary Debulking Gynaecological Surgery
Brief Title: The Effects of Hemodilution Methods in Patients Undergoing Primary Debulking Gynaecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhou Huidan, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-2015-194
Record Dates: First submitted 2023-09-23; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Neoplasm Epithelial
Keywords: Acute normovolemic hemodilution (ANH); Acute hypervolemic hemodilution (AHH); Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): In control group ，patients had undergone similar surgical and anesthesia procedures in the same time period but whose hemodynamic management was carried out according to the clinical decision of the attending anesthesiologist.
- acute normovolemic hemodilution (ANH) (Other): Before anesthesia induction, in the ANH Group, blood was withdrawn at a speed of 25-30ml/min from radial artery and stored in standard collection bags. The volume of blood to be removed during ANH was calculated using an established formula as follows: V = EBV (H0 - Ht) / H. During collection, a tilt rocker scale was used to rock, mix, and weigh the blood. To maintain euvolemia, half of the blood volume removed was replaced with 6% hydroxyethyl starch 130/0.4 with medium molecular weight at a 1:1 ratio and half was replaced with crystalloid at a 1:2 ratio. The autologous blood was returned to patients if the intraoperative transfusion trigger (Hb <8.0g/dl) was reached or at the completion of the operation.
  Interventions: Other: acute normovolemic hemodilution (ANH)
- acute hypervolemic hemodilution (AHH) (Other): In AHH group, 15ml/kg Voluven was transfused at a speed of 30 ml/min to make Hct to drop to medium. In control group, the regular transfusion and infusion were conducted. Allogenic blood was only given after all autologous blood had been returned to the patient. The transfusion triggers (Hb <8.0g/dl) were used to determine the need for allogenic blood transfusions during the procedure in three groups.
  Interventions: Other: acute hypervolemic hemodilution (AHH)

INTERVENTIONS:
Other: acute normovolemic hemodilution (ANH) — Acute normovolemic hemodilution (ANH) is a medical procedure that involves removing a certain volume of blood from a patient before surgery and replacing it with a volume expander or blood substitute. The goal of ANH is to reduce the need for blood transfusions during or after surgery. During the ANH procedure, a patient's blood is typically withdrawn and replaced with a crystalloid or colloid solution. This dilutes the patient's blood, reducing the concentration of red blood cells. The withdrawn blood is then stored and can be reinfused back into the patient after the surgical procedure is completed.
  Arms: acute normovolemic hemodilution (ANH)
Other: acute hypervolemic hemodilution (AHH) — The purpose of diluting the blood with fluids and removing some of the red blood cells is to decrease the viscosity of the blood. This can improve blood flow and oxygen delivery to tissues, especially in cases of decreased blood flow or oxygenation.
  Arms: acute hypervolemic hemodilution (AHH)

SUMMARY:
Primary cytoreductive surgery for ovarian cancer is an ideal setting to evaluate endothelial function under ANH and AHH, as the procedure is associated with moderately high blood loss. As the technique has not yet been described in this setting, investigators designed a pilot study to evaluate ANH and AHH in patients planned to undergo primary cytoreduction during perioperative period, with the intent of proceeding to a randomized trial if results were favorable.

DETAILED DESCRIPTION:
Using a computer-generated random number table, patients were randomized to three groups: Control Group(n=30), ANH Group(n=30) and AHH Group(n=30). Patients underwent standard preoperative preparation for cytoreductive surgery according to institutional standards.All patients who underwent a standard anesthesia protocol and similar surgical procedures were considered for the analysis. For this purpose, investigators only included patients who underwent the following interventions: radical hysterectomy, bilateral adnexectomy, one or more bowel resection, peritonectomy, pelvic lymphadenectomy and extended periaortic lymphadenectomy. The patient would be ruled out of the experiment when the participant was accompanied with any kind of serious complications such as wakening delay and drug allergy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of advanced primary epithelial ovarian
2. No comorbidities nor functional limitations (ASA Grade II due to high tumor load)
3. Serum hemoglobin (Hb) before surgery ≥ 11g/dl
4. Hematocrit (Hct) ≥ 35%
5. Quantity of platelets ≥ 100 × 109 /L

Exclusion Criteria:

1. Age <18 or >65 years
2. Body mass index <20 and >30 kg/m2
3. Duration of surgery <180 min
4. Severe cardiovascular disease, liver and kidney disease
5. Thromboembolism history

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Endothelin-1 (ET-1) | three periods: before hemodilution, immediate postoperative period, and 24 hours later
  Blood sample (5 ml) was obtained from the vein，Endothelin-1 (ET-1) was measured using the enzyme-linked immunosorbent assay (ELISA) (Merck & Co Inc, USA) according to manufacturer's instructions.

SECONDARY OUTCOMES:
von Willebrand factor (VWF), tissue factor pathway inhibitor (TFPI), plasminogen activator inhibitor 1 (PAI-1) and thrombomodulin (TM) levels | three periods: before hemodilution, immediate postoperative period, and 24 hours later
  von Willebrand factor (VWF), tissue factor pathway inhibitor (TFPI), plasminogen activator inhibitor 1 (PAI-1) and thrombomodulin (TM) levels were measured using the enzyme-linked immunosorbent assay (ELISA) (Merck & Co Inc, USA) according to manufacturer's instructions.